CLINICAL TRIAL: NCT01586585
Title: Patient Rehabilitation Post Cardiac Surgery Based on Their Pre-op Status
Brief Title: Back to Functional Life Following Cardiac Surgery
Acronym: BTFL2012
Status: Withdrawn | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-12-0021-CTIL
Record Dates: First submitted 2012-04-22; First posted 2012-04-27 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Cardiac Study Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- post cardiac surgery patients

SUMMARY:
The investigators will monitor cardiac patients rehabilitation post op upon their pre op status.

DETAILED DESCRIPTION:
In this work we will try to monitor the patients for a longer period, starting from their hospitalization period through their rehabilitation period up to 18 months post their discharge from the hospital.

Many studies tried to evaluate different ways to predict postoperative complications following cardiac surgery, patient's survival, rehabilitation rate and duration. Today, following these studies doctors use different methods to evaluate these parameters. The Society of Thoracic Surgeons mortality risk score (STS) and the European System for Cardiac Operative Risk Evaluation (EuroSCORE) scoring system are the two most frequently used risk profile systems within the United States and Europe. The STS score is comprised of over 40 clinical parameters, whereas the EuroSCORE involves 18 clinical characteristics that comprises three categories, each weighted accordingly. Studies published recently suggest that a combination of a new frailty score and the traditional scoring systems may facilitate a more accurate risk scoring in elderly high-risk patients scheduled for conventional cardiac surgery or trans-catheter aortic valve replacement.

In this study we will try to evaluate the contribution of using a frailty score index in addition to the EuroSCORE evaluation in patients≥50 years of age, in prediction of postoperative complications following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing cardiothoracic surgery in the Cardiothoracic Surgery Department at Carmel Medical center, Haifa, Israel, between: 1.5.12-28.2.14.
2. Patients ≥ 50 years of age
3. Informed consent from each participant that can understand, read and sign the informed consent form.

Exclusion Criteria:

1. Emergent surgery, defined as a surgery for which there should be no delay due to ongoing refractory cardiac compromise.
2. Clinical instability, defined as active coronary ischemia, decompensated heart failure not yet stabilized, or any acute process causing significant symptoms or abnormal vital signs.
3. Severe neuropsychiatric condition causing inability to cooperate with the study procedures.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Length of time taken to the patient to get back to functional life | 3 years
  The back to functional life period will be estimated using questionnaires that will be filled by the patient before the operation and in intervals after the operation

SECONDARY OUTCOMES:
Number of Participants with Adverse Events stratified by Frailty index | 3 years
  The patients will go through different tests in order to estimate their fragility index, their post op complications will be monitored, and we will try to find association between the frailty index and severity and number of complications

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Barac, MD/PhD, Principal Investigator — Cramel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel